CLINICAL TRIAL: NCT05981274
Title: A Prospective and Retrospective Interventional Study on the Bone-health Effectiveness of Applying Recombinant Factor VIII Fc (rFVIIIFc) to Patients With Hemophilia A (Prototype A)
Brief Title: A Study on the Bone-health Effectiveness of Applying Recombinant Factor VIII Fc (rFVIIIFc) to Patients With Hemophilia A (Prototype A)
Status: Recruiting | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chen Yeu-Chin, Director of the Hemophilia Center, Tri-Service General Hospital
Other Study IDs: A202305097
Record Dates: First submitted 2023-07-17; First posted 2023-08-08 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-07

CONDITIONS: Severe Hemophilia A Without Inhibitor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples (serum) will be obtained for serum markers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Systematic joint and bone health assessments before and after enrollment: 1. Haemophilia Early Arthropathy Detection :HEAD-US, HJHS, and DEXA scan
  2. serum markers : CTX-II, COMP, hsCRP, TNF-a, CTX-I, sRANKL, OPG, and Osteopontin (OPN)
  3. Quality of life assessments (Haem-A-QoL, EQ-5D)
  Interventions: Diagnostic Test: serum biomarker.

INTERVENTIONS:
Diagnostic Test: serum biomarker. — serum biomarker:CTX-II, COMP, hsCRP, TNF-a, CTX-I, sRANKL, OPG, and Osteopontin (OPN)

SUMMARY:
Study Objectives*

1. Provide a systematic evaluation of the treatment outcomes in patients with hemophilia A
2. Emphasize the importance and clinical benefits of rFVIII-Fc in joint and bone health.
3. Compare the clinical outcomes from 1 year before and after switching to EHL.
4. Exploratory: Identify biomarkers that could provide more useful and convenient evaluations of joint and bone health. (Time-saving and easy to monitor)

DETAILED DESCRIPTION:
In this study, we would like to focus on the evaluation of joint and bone health in persons with severe hemophilia A (PwHA) treated with rFVIIIFc prophylaxis. We also aim to identify potential biomarkers for assessing the joint and bone health of PwHA. Since the joint and bone health examinations are time-consuming, expensive, and require special equipment, the patients could only receive the examinations annually to realize the status of their joint health. The biomarkers testing will provide a more convenient and time-saving option on the joint and bone health evaluation for PwHA. Therefore, surrogate of biochemical marker(s) to represent the joint and BMD progression is an unmet need for clinical practice. Investigating different biomarkers and combining them with the joint and BMD results to provide a systematic approach for elucidating the treatment outcomes of PwHA treated with rFVIIIFc is major goal of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe hemophilia A (all ages).
2. Patients with moderate type hemophilia A with hemophilic arthropathy.
3. Currently on rFVIIIFc regular prophylaxis and have previous medical record with regular prophylaxis with standard half-life product for one year
4. Able and willing to undergo joint and bone examinations

Exclusion Criteria:

1. Participants of other interventional studies.
2. Patients with current inhibitors.
3. History of major neurological disease (eg. Stroke, Parkinson's disease, neuropathy, etc.)
4. History of major psychiatric disease (eg. Schizophrenia, bipolar disorder)
5. Significantly impaired vision/hearing

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Males with one affected X chromosome is defined hemophilia disease; a female with one affected X chromosome is a "carrier" of hemophilia.
Study Population: severe hemophilia A patients or moderate hemophilia A patients with hemophilic arthropathy.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Systematic joint and bone health assessments before and after enrollment | up to 5 years
  Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) on patients' ankles, knees, and elbows. Also evaluate the Hemophilia Joint Health Score (HJHS) and Dexa scan at the hip.

SECONDARY OUTCOMES:
Serum markers | up to 5 years
  CTX-II, COMP, HSCRP, TNF-ALPHA, CTX-I, SRANKL, OPG, OPN

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital Hemophilia Care Center, Taipei, Neihu Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No